CLINICAL TRIAL: NCT01763255
Title: The Safety of Multiple Intrathecal Injection of Bone Marrow Derived CD133 Cells in Patients With Cerebral Palsy
Brief Title: Multiple Transplantation of Bone Marrow Derived CD133 Cell in Cerebral Palsy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Royan Institute (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Royan-Nerve-003
Record Dates: First submitted 2012-12-25; First posted 2013-01-08 (Estimated); Last update posted 2014-04-25 (Estimated); Status verified 2011-01

CONDITIONS: Cerebral Palsy
Keywords: cerebral palsy CD133 cells intrathecal injection
MeSH Terms: conditions — Cerebral Palsy | interventions — Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CD133 transplantation (Experimental): The patients with cerebral palsy that underwent CD133 transplantation.
  Interventions: Biological: stem cell intrathecal injection
- Control (No Intervention): The patients with cerebral palsy that underwent regular observation.

INTERVENTIONS:
Biological: stem cell intrathecal injection — Intrathecal injection of Bone marrow derived CD133 cells
  Other Names: Stem cell transplantation
  Arms: CD133 transplantation

SUMMARY:
Cerebral palsy (CP) is condition, sometimes thought of as a group of disorders that can involve brain and nervous system functions such as movement, learning, hearing, seeing, and thinking.Cerebral palsy is caused by injuries or abnormalities of the brain. Most of these problems occur as the baby grows in the womb, but they can happen at any time during the first 2 years of life, while the baby's brain is still developing.Bone marrow derived stem cells are known as a effective therapy.

In this study the investigators evaluate the side effect of multiple intrathecal injection of bone marrow stem cell in patients with cerebral palsy.

DETAILED DESCRIPTION:
In this study,we evaluate the safety of multiple transplantation of bone marrow derived stem cells.the children(4-12years)with definite diagnose of cerebral palsy enroll to the study.first of all all the physical exam,laboratory test,EEG and MRI is done.after hospital admission,the patient underwent bone marrow transplantation.In laboratory,the cells are separated and prepared for injection.after 24hours the neurosurgeon inject the cells(intrathecal).the patient would be under observed for 48hours.If no allergic reaction or abnormal neurological symptoms accrued,patients can be discharged and would be followed up 1,3 and 6months after injection.at the end of the 6months,the patients would receive second injection as same as the previous process.then they are followed at 1,3 immediate local and systemic side effect(fever,respiratory distress,erythema,rash,increase of heart rate or blood pressure)and neurological symptoms:motor dysfunction,sensory dysfunction,sphincter dysfunction,nausea,vomiting,head ache.EEG,MRI,GMFM66

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of spastic quadriplegic CP Children must be between the ages of 4 and 12 years Children must be cleared by an orthopedic surgeon for risk of hip subluxation or dislocation and cannot have significant scoliosis (curvature > 40 degrees) Children must be seizure-free or seizure controlled

Exclusion Criteria:

* Children who have a diagnosis of "mixed" types of CP (i.e. athetosis) or other movement disorders (i.e. ataxia) Children who have had a selective dorsal rhizotomy, are presently are receiving intrathecal Baclofen, or have changed their spasticity medications in the past 6 months.

Children who have a metallic or electrical implants

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 8 (Actual)
Dates: Start 2012-04; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
motor dysfunction | 6months
  Evaluation the motor dysfunction 6months after intrathecal injection.
sensory dysfunction | 6months
  Evaluation the sensory dysfunction after intrathecal injection of CD133 cells.
unconsciousness | 48hours
  Evaluation the rate of unconsciousness during 48hours after cell transplantation.
fever | 48hours
  Evaluation the symptom of infection like fever 48hours after cell transplantation.

SECONDARY OUTCOMES:
motor improvement | 6months
  Measure the improvement of motor system by GMFM66.
Balance improvement | 6months
  Measure the balance improvement by BBS.
Spasm | 6months
  Evaluation the improvement of spasm after stem cell transplantation.

CONTACTS AND LOCATIONS:
Overall Officials: Hamid Gourabi, PhD, Study Chair — Head of Royan Institute; Nasser Aghdami, MD,PhD, Study Director — Head of Royan department of degenerative medicine,Head of Royan celltherapy center; Ali Reza Zali, MD, Study Director — Head of Neurosurgery research center of Shahid Beheshti University
Locations (1):
- Royan Institute, Tehran, Iran

REFERENCES:
- See also: Related Info — http://Royaninstitute.org